CLINICAL TRIAL: NCT00264771
Title: The Hospital Based Incidence of Acute Rheumatic Fever and Rheumatic Heart Disease, Acute Post Streptococcal Glomerulonephritis and Invasive Group A Streptococcal Disease in Fiji
Brief Title: Hospital Based Incidence of Group A Streptococcal Disease in Fiji
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0082
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2007-10

CONDITIONS: Streptococcus Group A
Keywords: Fiji, Group A streptococcus, rheumatic, glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this ongoing study (Part II) is to estimate the incidence of acute rheumatic fever, rheumatic heart disease, acute post-streptococcal glomerulonephritis (kidney disease), and invasive group A streptococcal (GAS) disease (strep infection) in Fiji to help develop better treatments and vaccines. Group A streptococcal disease is caused by the bacterium group A streptococcus. It is commonly found in the nose and throat of normal healthy adults and children, and can cause illness. The bacterium is spread by close contact with patients or carriers, through things like coughing, sneezing, kissing, or sharing a drink and can cause a wide variety of illnesses. These illnesses may be a sore throat, skin sores, and less commonly acute rheumatic fever or kidney disease. Participants of all ages will be recruited through the Colonial War Memorial and Lautoka Hospital. A blood sample will be collected from each study participant. Subject participation should be less than one day.

DETAILED DESCRIPTION:
This study is a prospective active surveillance study of group A streptococcal (GAS) diseases across two hospital sites designed to estimate the local incidence of acute rheumatic fever (ARF), rheumatic heart disease (RHD), acute post streptococcal glomerulonephritis (APSGN) and invasive GAS disease. It is part II of a series of 5 studies including DMID protocols 05-0081, 05-0117, 05-0118, and 06-0081. The study is also designed to assess the clinical features of these GAS diseases. The study will also provide detailed information about the molecular epidemiology of GAS from these diseases. The study will establish an active surveillance system for cases of ARF and APSGN and invasive GAS disease at the Colonial War Hospital, in Suva Fiji and at Lautoka Hospital, Lautoka. In addition, the study will establish an active surveillance system for patients presenting with complications of established RHD at the Colonial War Memorial Hospital in Suva Fiji. The primary objectives of the study are to estimate the incidence of: acute rheumatic fever in the Western and Central divisions of Fiji in children 3-17 years of age and adults 18-40 years; RHD in all ages in the Central division of Fiji; APSGN in the Western and Central divisions of Fiji in children 0-17 years of age; and invasive GAS disease in the Western and Central divisions of Fiji in all ages. The secondary objectives of the study are to: describe the clinical features of patients presenting with complications of established RHD in the central division of Fiji; establish an ongoing surveillance system for GAS diseases in the Western and Central divisions; describe the clinical features of patients presenting with ARF, APSGN and invasive GAS disease in Fiji; genotypically characterize GAS isolates from patients with ARF, APSGN and invasive GAS disease in Fiji; and measure anti-J8 antibodies in patients with GAS disease. The primary endpoints of the study are to determine the incidence of: confirmed and probable ARF, both first presentation and recurrent cases; RHD in all ages in the Central division of Fiji; confirmed and probable APSGN; and confirmed and probable invasive GAS disease. The secondary endpoints of the study include: incidence of heart failure, atrial fibrillation, stroke and infective endocarditis in patients with RHD presenting to Colonial War Memorial Hospital; distribution of symptoms and signs of ARF in patients presenting to hospital with ARF; distribution of sites of infection in cases of invasive GAS disease; incidence of necrotizing fasciitis and streptococcal toxic shock syndrome; proportion of GAS isolates from patients with ARF, APSGN and invasive GAS disease that contain the J8 epitope and the overall emm-type distribution of GAS isolates; characterization of GAS isolates (C repeat region sequencing and emm-typing); and measurement of anti-J8 antibodies in patients with GAS disease.

ELIGIBILITY:
Inclusion Criteria:

Informed consent will be obtained from all study participants. Children between 0 -17 years of age will be enrolled in the APSGN study. Children between 3-17 years of age and adults between 18-40 years will be enrolled in the ARF study. Children and adults of all ages will be enrolled in the RHD and invasive GAS studies.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550
Dates: Start 2005-12; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Locations (2):
- Fiji (2):
  - Lautoka Hospital, Lautoka
  - Colonial War Memorial Hospital, Suva